CLINICAL TRIAL: NCT02133456
Title: A Post-marketing Safety Study of SIBP's Inactivated, Split-virion Influenza Vaccine Administered in Chinese Subjects Aged 3 Years and Older
Brief Title: A Post-marketing Safety Study of Inactivated, Split-virion Influenza Vaccine in Subjects Aged 3 Years and Older
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Principal Investigator, Wu Jiang, Department of Immunization and Prevention,Beijing Centers for Disease Control and Prevention, Centers for Disease Control and Prevention, China
Other Study IDs: BJCDCWJ201401
Record Dates: First submitted 2014-05-07; First posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Influenza; Vaccination Adverse Event
Keywords: safety; influenza vaccine; post-marketing
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Ecologic or Community
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- SIBP's vaccine: SIBP's vaccine group is the population injected with this vaccine.

SUMMARY:
To monitor the safety of Shanghai Institute of Biological Products Company's influenza vaccine in subjects aged 3 years and older through Adverse Events Following Immunization Surveillance System of China.

The hypothesis is that there is no significant difference in the occurrence of adverse events among influenza vaccines manufactured by SIBP and other companies.

DETAILED DESCRIPTION:
Inactivated split-virion vaccines from Shanghai Institute of Biological Products Company have been used for more than 10 years in Beijing population. Some 160 thousands doses have been sold to subjects aged 3 years and older in this area. We review and summarize spontaneously reported adverse events from safety surveillance.

Adverse events were collected through the Adverse Events Following Immunization (AEFI) Surveillance System. Beijing CDC and local prefectural CDC must organize an expert panel to investigate adverse events and assess causality, using criteria based on Chinese Standard Procedures for Vaccination. The panels consist of physicians, epidemiologists, pharmacists, and other relevant experts. In general, expert panels investigate deaths, life-threatening illnesses, and permanent disabilities, and immunization-program managers or vaccination providers investigate common, minor adverse events. Adverse events are classified into one of five categories: vaccine reactions (common and minor to rare and more serious), program errors, coincidental illnesses, psychogenic reactions, and unclassifiable events.

At the time of vaccination, vaccinees were instructed to report any adverse event to physicians or vaccination providers. The following adverse events were required to be reported: adverse events that were fatal or that resulted in disability and clusters of events (i.e., notably high numbers of similar adverse events related to a certain vaccine) ; anaphylaxis or other allergic reactions occurring within 24 hours after vaccination; fever (axillary temperature, >37.5°C), angioedema, or a local injection-site reaction (diameter, >2.5 cm) occurring within 5 days after vaccination; purpura, an Arthus reaction, febrile convulsion, seizure, or polyneuritis occurring within 15 days after vaccination; and the Guillain-Barré syndrome occurring within 3 months after vaccination. Other reactions that were common and minor (e.g., mild pain and fatigue) were not required to be reported.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 3 years and above on the day of immunization, who are eligible for seasonal influenza vaccination.
* Recipients of SIBP's inactivated, split-virion influenza vaccine.

Exclusion Criteria:

* History of any serious reaction to flu vaccine, or any materials in the vaccine, and to eggs (including ovalbumin) and chicken protein.
* Receipt of a live vaccine within 4 weeks prior to Study Day 1.
* Any condition, which in the opinion of the study doctor, might interfere with the evaluation of the study objective.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Beijing subjects aged 3 years or older, at the time of routine visit to a participating clinic or hospital for influenza vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 166240 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
the rate of reported adverse events | 3 months after vaccination
  The rate of reported adverse events was calculated by dividing the number of vaccinees who reported having an event by the number of vaccine doses administered.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wu, Master, Principal Investigator — Beijing Centers for Disease Prevention and Control, China